CLINICAL TRIAL: NCT00000620
Title: Action to Control Cardiovascular Risk in Diabetes (ACCORD)
Acronym: ACCORD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute on Aging (NIA) (NIH); National Eye Institute (NEI) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 123; N01HC95178 (NIH); N01HC95179 (NIH); N01HC95180 (NIH); N01HC95181 (NIH); N01HC95182 (NIH); N01HC95183 (NIH); N01HC95184 (NIH); IAA#Y1HC9035 (Other Grant/Funding Number: U.S. Centers for Disease Control); IAA#Y1HC1010 (Other Grant/Funding Number: U.S. Centers for Disease Control); NCT00182910 (obsolete NCT alias)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2014-11

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus; Coronary Disease
Keywords: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus; Coronary Disease | interventions — glimepiride; Metformin; repaglinide; Rosiglitazone; Pioglitazone; Insulin; Isophane Insulin, Human; Insulin Aspart; Insulin Detemir; Insulin Glargine; Acarbose; Antihypertensive Agents; benazepril; Lisinopril; Ramipril; Chlorthalidone; Metoprolol; Diltiazem; Felodipine; Terazosin; candesartan; candesartan cilexetil; Valsartan; Furosemide; Reserpine; Hydralazine; Carvedilol; Triamterene; Hydrochlorothiazide; hydrochlorothiazide-triamterene; hydrochlorothiazide, lisinopril drug combination; Amlodipine; Simvastatin; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Glycemia Trial: intensive control (Experimental): Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%.
  Interventions: Drug: Anti-hyperglycemic Agents
- Glycemia Trial: standard control (Active Comparator): Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 - 7.9%.
  Interventions: Drug: Anti-hyperglycemic Agents
- BP Trial: intensive control (Experimental): Open label administration of anti-hypertensive agents to reduce and maintain systolic blood pressure (SBP) level to <120 mmHg.
  Interventions: Drug: Anti-hypertensive Agents
- BP Trial: standard control (Active Comparator): Open label administration of multiple anti-hypertensive agents to maintain SBP level <140 mm Hg.
  Interventions: Drug: Anti-hypertensive Agents
- Lipid Trial: fenofibrate (Experimental): Double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m2 in combination with open label simvastatin.
  Interventions: Drug: Blinded fenofibrate or placebo plus simvastatin
- Lipid Trial: placebo (Placebo Comparator): Double blind administration of placebo matching either 160 mg/day in participants with eGFR ≥50 mL/min/1.73m2 or 54 mg/day in participants with eGFR <50 mL/min/1.73m2 in combination with open label simvastatin.
  Interventions: Drug: Blinded fenofibrate or placebo plus simvastatin

INTERVENTIONS:
Drug: Anti-hyperglycemic Agents — Multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals (intensive control <6%; standard control 7.0-7.9%).
  Other Names: glimepiride (Amaryl); metformin (Glucophage); repaglinide (Gluconorm, Prandin); rosiglitazone (Avandia); pioglitazone (Actos); human regular insulin (Novolin ge Toronto); human NPH (Novolin N); human mixed (Novolin 70/30); human isophane (Novolin ge NPH); human 30/70 (Novolin ge 30/70); insulin aspart (NovoRapid, NovoLog); insulin detemir (Levemir); human regular insulin (Novolin R); insulin glargine (Lantus); Acarbose
  Arms: Glycemia Trial: intensive control; Glycemia Trial: standard control
Drug: Anti-hypertensive Agents — Multiple anti-hypertensive agents as needed to reach Blood Pressure Trial arm-specific goals (intensive control <120 mm Hg; standard control <140 mm Hg).
  Other Names: benazepril (Lotensin, Zestril, Altace); chlorthalidone (Thalitone); metoprolol (Toprol XL); diltiazem (Tiazac); plendil (Felodipine); terazosin (Hytrin); candesartan (Atacand); valsartan (Diovan); furosemide; reserpine; hydralazine; carvedilol (Coreg); triamterene / hydrochlorothiazide (Dyazide); metoprolol / hydrochlorothiazide(Lopressor HCT); benazepril / hydrochlorothiazide (Lotensin HCT); lisinopril / hydrochlorothiazide (Zestoretic); candesartan / hydrochlorothiazide (Atacand HCT); valsartan / hydrochlorothiazide (Diovan HCT); amlodipine / benazepril (Lotrel)
  Arms: BP Trial: intensive control; BP Trial: standard control
Drug: Blinded fenofibrate or placebo plus simvastatin — Double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m2 or matching placebo in combination with open label simvastatin 20 - 40 mg/day.
  Other Names: fenofibrate (Tricor)
  Arms: Lipid Trial: fenofibrate; Lipid Trial: placebo

SUMMARY:
The purpose of this study is to prevent major cardiovascular events (heart attack, stroke, or cardiovascular death) in adults with type 2 diabetes mellitus using intensive glycemic control, intensive blood pressure control, and multiple lipid management.

DETAILED DESCRIPTION:
BACKGROUND:

Currently, about 17 million Americans have been diagnosed with diabetes and more than 90 percent of them have type 2 diabetes. The number of people with this form of diabetes, formerly known as adult onset or non-insulin dependent diabetes, is growing rapidly. By 2050, the number of Americans with diagnosed diabetes is projected to increase by 165 percent to 29 million, of whom 27 million will have the type 2 form. Cardiovascular disease (CVD) is the leading cause of death in people with type 2 diabetes; these individuals die of CVD at rates two to four times higher than those who do not have diabetes. They also experience more nonfatal heart attacks and strokes.

Type 2 diabetes is associated with older age and is more common in those who are overweight or obese and have a family history of diabetes. Women with a history of diabetes during pregnancy, adults with impaired glucose tolerance, people with a sedentary lifestyle, and members of a minority race/ethnicity are also at a greater risk for developing type 2 diabetes. African Americans, Hispanic/Latino Americans, American Indians, and some Asian Americans and Pacific Islanders are at particularly high risk for type 2 diabetes.

DESIGN NARRATIVE:

The three strategies tested in ACCORD included the following: (1) Blood sugar - ACCORD was designed to determine whether lowering blood glucose to a level closer to normal than called for in current guidelines reduces CVD risk. The study estimated effects on CVD of that level compared with a level that is usually targeted. (2) Blood pressure - many people with type 2 diabetes have high blood pressure. The blood pressure part of the trial was designed to determine the effects of lowering blood pressure in the context of good blood sugar control, that is to determine whether lowering blood pressure to normal (systolic pressure less than 120 mm Hg) will better reduce CVD risk, as compared to a usually-targeted level in current clinical practice (i.e., below the definition of hypertension; systolic pressure less than 140 mm Hg). (3) Blood Fats - Many people with diabetes have high levels of LDL ("bad") cholesterol and triglycerides, as well as low levels of HDL ("good") cholesterol. ACCORD participants who are selected for this part of the trial were assigned to an intervention to improve blood fat levels. This part of the study looked at the effects of lowering LDL cholesterol and blood triglycerides and increasing HDL cholesterol compared to an intervention that only lowers LDL cholesterol, all in the context of good blood sugar control. A drug from a class of drugs called "fibrates" was used to lower triglycerides and increase HDL cholesterol, whereas a drug from the class of drugs called "statins" was used to lower LDL cholesterol.

All ACCORD participants received blood sugar treatment from the study. Based on the second trial (Blood Pressure or Lipid) they were assigned to, participants also received their high blood pressure or cholesterol care from the study. Study participants received all medication and treatments related to the study free of charge. Individuals who selected for and consented to participate in the ACCORD study continued to see their personal physician for all other health care.

In summary, the ACCORD Study was a double 2x2 factorial design with factors consisting of: intensive versus standard glycemic control, intensive versus standard blood pressure control, and blinded fenofibrate or placebo in combination with simvastatin to maintain desirable LDL-C levels. All 10,251 participants were randomized to the glycemic interventions; a subgroup of 4,733 participants who met the blood pressure entry criteria were randomized to the blood pressure interventions in one 2x2 trial; and a distinct subgroup of 5,518 participants who met the lipid entry criteria were randomized to the lipid interventions in the second 2x2 trial. All participants had established type 2 diabetes and were recruited from 77 clinical centers in the United States (64 sites) and Canada (13 sites).

On February 6, 2008, the National Heart, Lung and Blood Institute (NHLBI) announced that participants in the intensive glycemia treatment would be transitioned to the ACCORD standard glycemic treatment approach due to higher mortality in the intensive treatment group terminating the experimental arm of the Glycemia Trial early. The Blood Pressure and Lipid trials continued as designed to their planned termination in 2009.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus, as determined by the new American Diabetes Association guidelines, which include a fasting plasma glucose level greater than 126 mg/dl (7.0 mmol/l), or a 2-hour postload value in the oral glucose tolerance test of greater than 200 mg/dl, with confirmation by a retest
* For participants aged 40 years or older, history of CVD (heart attack, stroke, history of coronary revascularization, history of peripheral or carotid revascularization, or demonstrated angina)
* For participants aged 55 years or older, a history of CVD is not required, but participant must be considered to be at high risk for experiencing a CVD event due to existing CVD, subclinical disease, or 2+ CVD risk factors
* HbA1c 7.5%-9% (if on more drugs) or 7.5%-11% (if on fewer drugs)

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10251 (Actual)
Dates: Start 1999-09; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Simons-Morton, MD, PhD, Study Director — National Heart, Lung, and Blood Institute (NHLBI); William Friedewald, MD, Study Chair — Columbia University, New York, NY; Robert Byington, PhD, Principal Investigator — Wake Forest University, Winston-Salem, NC
Locations (7):
- United States (6):
  - Minneapolis Medical Research Foundation, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Veterans Affairs, Memphis, Tennessee
  - University of Washington, Seattle, Washington
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Cushman WC, Grimm RH Jr, Cutler JA, Evans GW, Capes S, Corson MA, Sadler LS, Alderman MH, Peterson K, Bertoni A, Basile JN; ACCORD Study Group. Rationale and design for the blood pressure intervention of the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):44i-55i. doi: 10.1016/j.amjcard.2007.03.005. Epub 2007 Apr 16. PMID 17599425
- [Background] Williamson JD, Miller ME, Bryan RN, Lazar RM, Coker LH, Johnson J, Cukierman T, Horowitz KR, Murray A, Launer LJ; ACCORD Study Group. The Action to Control Cardiovascular Risk in Diabetes Memory in Diabetes Study (ACCORD-MIND): rationale, design, and methods. Am J Cardiol. 2007 Jun 18;99(12A):112i-122i. doi: 10.1016/j.amjcard.2007.03.029. Epub 2007 Apr 12. PMID 17599421
- [Background] Sullivan MD, Anderson RT, Aron D, Atkinson HH, Bastien A, Chen GJ, Feeney P, Gafni A, Hwang W, Katz LA, Narayan KM, Nwachuku C, O'Connor PJ, Zhang P; ACCORD Study Group. Health-related quality of life and cost-effectiveness components of the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial: rationale and design. Am J Cardiol. 2007 Jun 18;99(12A):90i-102i. doi: 10.1016/j.amjcard.2007.03.027. Epub 2007 Apr 13. PMID 17599429
- [Background] Bonds DE, Kurashige EM, Bergenstal R, Brillon D, Domanski M, Felicetta JV, Fonseca VA, Hall K, Hramiak I, Miller ME, Osei K, Simons-Morton DG; ACCORD Study Group. Severe hypoglycemia monitoring and risk management procedures in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):80i-89i. doi: 10.1016/j.amjcard.2007.03.026. Epub 2007 Apr 17. PMID 17599428
- [Background] Kingry C, Bastien A, Booth G, Geraci TS, Kirpach BR, Lovato LC, Margolis KL, Rosenberg Y, Sperl-Hillen JM, Vargo L, Williamson JD, Probstfield JL; ACCORD Study Group. Recruitment strategies in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):68i-79i. doi: 10.1016/j.amjcard.2007.03.025. Epub 2007 Apr 12. PMID 17599427
- [Background] Ginsberg HN, Bonds DE, Lovato LC, Crouse JR, Elam MB, Linz PE, O'connor PJ, Leiter LA, Weiss D, Lipkin E, Fleg JL; ACCORD Study Group. Evolution of the lipid trial protocol of the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):56i-67i. doi: 10.1016/j.amjcard.2007.03.024. Epub 2007 Apr 12. PMID 17599426
- [Background] Goff DC Jr, Gerstein HC, Ginsberg HN, Cushman WC, Margolis KL, Byington RP, Buse JB, Genuth S, Probstfield JL, Simons-Morton DG; ACCORD Study Group. Prevention of cardiovascular disease in persons with type 2 diabetes mellitus: current knowledge and rationale for the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):4i-20i. doi: 10.1016/j.amjcard.2007.03.002. Epub 2007 Apr 12. PMID 17599424
- [Background] Gerstein HC, Riddle MC, Kendall DM, Cohen RM, Goland R, Feinglos MN, Kirk JK, Hamilton BP, Ismail-Beigi F, Feeney P; ACCORD Study Group. Glycemia treatment strategies in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Am J Cardiol. 2007 Jun 18;99(12A):34i-43i. doi: 10.1016/j.amjcard.2007.03.004. Epub 2007 Apr 19. PMID 17599423
- [Background] ACCORD Study Group; Buse JB, Bigger JT, Byington RP, Cooper LS, Cushman WC, Friedewald WT, Genuth S, Gerstein HC, Ginsberg HN, Goff DC Jr, Grimm RH Jr, Margolis KL, Probstfield JL, Simons-Morton DG, Sullivan MD. Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial: design and methods. Am J Cardiol. 2007 Jun 18;99(12A):21i-33i. doi: 10.1016/j.amjcard.2007.03.003. Epub 2007 Apr 16. PMID 17599422
- [Background] Chew EY, Ambrosius WT, Howard LT, Greven CM, Johnson S, Danis RP, Davis MD, Genuth S, Domanski M; ACCORD Study Group. Rationale, design, and methods of the Action to Control Cardiovascular Risk in Diabetes Eye Study (ACCORD-EYE). Am J Cardiol. 2007 Jun 18;99(12A):103i-111i. doi: 10.1016/j.amjcard.2007.03.028. Epub 2007 Apr 13. PMID 17599420
- [Result] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Derived] Liu M, Pei J, Zeng C, Xin Y, Tang P, Tang L, Hu X. BRI shows stronger association than BMI for MACE in patients with T2DM: insights from the ACCORD study. Front Nutr. 2025 Dec 12;12:1720948. doi: 10.3389/fnut.2025.1720948. eCollection 2025. PMID 41459091
- [Derived] Liu M, Pei J, Zeng C, Xin Y, Tang P, Hu X. Associations and predictive value of weight-adjusted waist index for cardiovascular outcomes in type 2 diabetes: evidence from the ACCORD study. Nutr J. 2025 Dec 17;24(1):184. doi: 10.1186/s12937-025-01251-0. PMID 41408264
- [Derived] Lavallee SK, Carew AS, Warren RA, Sapp JL, Levy AP, Andreou P, Herman CR, Rimm EB, Cahill LE. Haptoglobin Phenotype and Cardiovascular Risk: The ACCORD Blood Pressure RCT. Hypertension. 2026 Jan;83(1):189-198. doi: 10.1161/HYPERTENSIONAHA.125.25021. Epub 2025 Nov 11. PMID 41216699
- [Derived] Sano Y, Jin R, Yoshioka H, Nakazato Y, Sato H, Hisaka A. Development of a Novel Machine Learning Method for Estimation of Life-Long Chronic Disease Progression and Its Application to Type 2 Diabetes. Clin Transl Sci. 2025 Oct;18(10):e70351. doi: 10.1111/cts.70351. PMID 41127917
- [Derived] Wang J, Lv W, Wang Z, Li S, Wang Z, Zhou L, Wang Y, Ren L, Jiang C, He L, Xia S, Kong X, Zuo S, Kong Y, Guo X, Liu X, Li S, Tang R, Long D, Sang C, Zhou N, Du X, Dong J, Ma C. Orthostatic Systolic Blood Pressure Elevation and Incident Atrial Fibrillation: Insights From the SPRINT Trial. J Clin Hypertens (Greenwich). 2025 Aug;27(8):e70122. doi: 10.1111/jch.70122. PMID 40845203
- [Derived] Wang Z, Wang J, He L, Jiang C, Wang Y, Shen T, Zhao M, Li E, Zhou N, Sang C, Du X, Dong J, Ma C. Intensive Blood Pressure Control in Patients With Diabetes and Previous Stroke: A Post-Hoc Analysis of ACCORD-BP Trial. J Clin Hypertens (Greenwich). 2025 Jul;27(7):e70095. doi: 10.1111/jch.70095. PMID 40685691
- [Derived] Liu M, Pei J, Zeng C, Xin Y, Tang P, Hu X. Association and predictive value of the triglyceride glucose-weight adjusted waist index for cardiovascular outcomes in patients with type 2 diabetes. Sci Rep. 2025 Jul 8;15(1):24573. doi: 10.1038/s41598-025-08580-4. PMID 40628839
- [Derived] Yang Y, Xing Z. Depressive Symptoms and Metabolic Dysregulation Control: A Closer Look at Control Challenges in T2DM Patients. Depress Anxiety. 2024 Sep 27;2024:7115559. doi: 10.1155/2024/7115559. eCollection 2024. PMID 40226732
- [Derived] Cheng Y, Zhu XB, Xu YL, Zou J, Huang W, Tian J, Sheng CS. Time in target range of systolic blood pressure and eGFR slope in patients with type 2 diabetes. Hypertens Res. 2025 May;48(5):1787-1798. doi: 10.1038/s41440-025-02173-4. Epub 2025 Mar 10. PMID 40065086
- [Derived] Li S, Lin L, Chen X, Liu S, Gao M, Cheng X, Li C. Association between body fat variation rate and risk of diabetic nephropathy - a posthoc analysis based on ACCORD database. BMC Public Health. 2024 Oct 14;24(1):2805. doi: 10.1186/s12889-024-20317-y. PMID 39396960
- [Derived] Zhang W, Huang Y, Zhou Z, Xie P, Zhuang X, Jiang J, Liao X. Cardiac autonomic neuropathy modified the association between obesity and hypoglycemia in type 2 diabetes. Endocrine. 2024 Sep;85(3):1213-1221. doi: 10.1007/s12020-024-03728-0. Epub 2024 Jun 21. PMID 38904908
- [Derived] Yang R, Jiang H, Xing Z, Ding H, Yin Z, Fu L, Tai S. Cumulative blood pressure predicts risk of stroke in individuals with type 2 diabetes. Diabetes Metab Syndr. 2024 Mar;18(3):102988. doi: 10.1016/j.dsx.2024.102988. Epub 2024 Mar 15. PMID 38513321
- [Derived] Zhou Y, Chai X, Yang G, Sun X, Xing Z. Changes in body mass index and waist circumference and heart failure in type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2023 Dec 21;14:1305839. doi: 10.3389/fendo.2023.1305839. eCollection 2023. PMID 38179309
- [Derived] Cromer SJ, Thaweethai T, Wexler DJ. Racial/ethnic and socioeconomic disparities in achievement of treatment goals within a clinical trial: a secondary analysis of the ACCORD trial. Diabetologia. 2023 Dec;66(12):2261-2274. doi: 10.1007/s00125-023-05997-2. Epub 2023 Sep 16. PMID 37715820
- [Derived] King JB, Berchie RO, Derington CG, Marcum ZA, Scharfstein DO, Greene TH, Herrick JS, Jacobs JA, Zheutlin AR, Bress AP, Cohen JB. New Users of Angiotensin II Receptor Blocker-Versus Angiotensin-Converting Enzyme Inhibitor-Based Antihypertensive Medication Regimens and Cardiovascular Disease Events: A Secondary Analysis of ACCORD-BP and SPRINT. J Am Heart Assoc. 2023 Sep 5;12(17):e030311. doi: 10.1161/JAHA.123.030311. Epub 2023 Aug 30. PMID 37646208
- [Derived] Kloecker DE, Davies MJ, Pitocco D, Khunti K, Zaccardi F. Intensive glucose control and recurrent cardiovascular events: 14-year follow-up investigation of the ACCORDION study. Diabetes Metab Res Rev. 2023 Jul;39(5):e3634. doi: 10.1002/dmrr.3634. Epub 2023 Apr 4. PMID 36905248
- [Derived] Zhou C, Zhang Y, Yang S, He P, Wu Q, Ye Z, Liu M, Zhang Y, Li R, Liu C, Jiang J, Hou FF, Nie J, Qin X. Associations between visceral adiposity index and incident nephropathy outcomes in diabetic patients: Insights from the ACCORD trial. Diabetes Metab Res Rev. 2023 Mar;39(3):e3602. doi: 10.1002/dmrr.3602. Epub 2022 Dec 30. PMID 36546623
- [Derived] Tang X, Zhu Y, Xing Z. Predicted lean body mass, fat mass, and heart failure in patients with type 2 diabetes mellitus. Am Heart J. 2023 Mar;257:78-84. doi: 10.1016/j.ahj.2022.12.008. Epub 2022 Dec 14. PMID 36528115
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Xing Z, Long C, Hu X, Chai X. Obesity is associated with greater cognitive function in patients with type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2022 Oct 24;13:953826. doi: 10.3389/fendo.2022.953826. eCollection 2022. PMID 36353230
- [Derived] Long C, Tang Y, Huang J, Liu S, Xing Z. Association of long-term visit-to-visit variability of HbA1c and fasting glycemia with hypoglycemia in type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2022 Aug 11;13:975468. doi: 10.3389/fendo.2022.975468. eCollection 2022. PMID 36034445
- [Derived] Tai S, Fu L, Zhang N, Yang R, Zhou Y, Xing Z, Wang Y, Zhou S. Association of the cumulative triglyceride-glucose index with major adverse cardiovascular events in patients with type 2 diabetes. Cardiovasc Diabetol. 2022 Aug 23;21(1):161. doi: 10.1186/s12933-022-01599-1. PMID 35999546
- [Derived] Fu L, Tai S, Sun J, Zhang N, Zhou Y, Xing Z, Wang Y, Zhou S. Remnant Cholesterol and Its Visit-to-Visit Variability Predict Cardiovascular Outcomes in Patients With Type 2 Diabetes: Findings From the ACCORD Cohort. Diabetes Care. 2022 Sep 1;45(9):2136-2143. doi: 10.2337/dc21-2511. PMID 35834242
- [Derived] Hukportie DN, Li FR, Zhou R, Zheng JZ, Wu XX, Zou MC, Wu XB. Lipid variability and risk of microvascular complications in Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial: A post hoc analysis. J Diabetes. 2022 Jun;14(6):365-376. doi: 10.1111/1753-0407.13273. Epub 2022 Jun 6. PMID 35668633
- [Derived] Hukportie DN, Li FR, Zhou R, Zheng JZ, Wu XX, Wu XB. Waist Circumference and Body Mass Index Variability and Incident Diabetic Microvascular Complications: A Post Hoc Analysis of ACCORD Trial. Diabetes Metab J. 2022 Sep;46(5):767-780. doi: 10.4093/dmj.2021.0258. Epub 2022 May 10. PMID 35584801
- [Derived] Tai S, Fu L, Zhang N, Zhou Y, Xing Z, Wang Y. Impact of Baseline and Trajectory of Triglyceride-Glucose Index on Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2022 Mar 24;13:858209. doi: 10.3389/fendo.2022.858209. eCollection 2022. PMID 35399955
- [Derived] Kaze AD, Jaar BG, Fonarow GC, Echouffo-Tcheugui JB. Diabetic kidney disease and risk of incident stroke among adults with type 2 diabetes. BMC Med. 2022 Mar 29;20(1):127. doi: 10.1186/s12916-022-02317-0. PMID 35346165
- [Derived] Sheng CS, Miao Y, Ding L, Cheng Y, Wang D, Yang Y, Tian J. Prognostic significance of visit-to-visit variability, and maximum and minimum LDL cholesterol in diabetes mellitus. Lipids Health Dis. 2022 Feb 10;21(1):19. doi: 10.1186/s12944-022-01628-8. PMID 35144636
- [Derived] Xing Z, Chai X. Changes in fat mass and lean body mass and outcomes in type 2 diabetes mellitus. Intern Emerg Med. 2022 Jun;17(4):1073-1080. doi: 10.1007/s11739-021-02916-4. Epub 2022 Feb 1. PMID 35106709
- [Derived] Kaze AD, Erqou S, Santhanam P, Bertoni AG, Ahima RS, Fonarow GC, Echouffo-Tcheugui JB. Variability of adiposity indices and incident heart failure among adults with type 2 diabetes. Cardiovasc Diabetol. 2022 Feb 1;21(1):16. doi: 10.1186/s12933-021-01440-1. PMID 35105339
- [Derived] Warren RA, Carew AS, Andreou P, Herman C, Levy AP, Ginsberg HN, Sapp J, Rimm EB, Kirkland S, Cahill LE. Haptoglobin Phenotype Modifies the Effect of Fenofibrate on Risk of Coronary Event: ACCORD Lipid Trial. Diabetes Care. 2022 Jan 1;45(1):241-250. doi: 10.2337/dc21-1429. PMID 34785535
- [Derived] Hukportie DN, Li FR, Zhou R, Zou MC, Wu XX, Wu XB. Association of Predicted Lean Body Mass and Fat Mass With Incident Diabetic Nephropathy in Participants With Type 2 Diabetes Mellitus: A Post Hoc Analysis of ACCORD Trial. Front Endocrinol (Lausanne). 2021 Oct 27;12:719666. doi: 10.3389/fendo.2021.719666. eCollection 2021. PMID 34777240
- [Derived] Gao S, Zhang H, Long C, Xing Z. Association Between Obesity and Microvascular Diseases in Patients With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Oct 26;12:719515. doi: 10.3389/fendo.2021.719515. eCollection 2021. PMID 34764938
- [Derived] Fu L, Zhou Y, Sun J, Zhu Z, Xing Z, Zhou S, Wang Y, Tai S. Atherogenic index of plasma is associated with major adverse cardiovascular events in patients with type 2 diabetes mellitus. Cardiovasc Diabetol. 2021 Oct 5;20(1):201. doi: 10.1186/s12933-021-01393-5. PMID 34610830
- [Derived] Shi S, Gouskova N, Najafzadeh M, Wei LJ, Kim DH. Intensive versus standard blood pressure control in type 2 diabetes: a restricted mean survival time analysis of a randomised controlled trial. BMJ Open. 2021 Sep 13;11(9):e050335. doi: 10.1136/bmjopen-2021-050335. PMID 34518266
- [Derived] Hukportie DN, Li FR, Zhou R, Zheng JZ, Wu XX, Wu XB. Anthropometric Measures and Incident Diabetic Nephropathy in Participants With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Aug 4;12:706845. doi: 10.3389/fendo.2021.706845. eCollection 2021. PMID 34421824
- [Derived] Ferreira JP, Ferrao D, Rossignol P, Zannad F, Sharma A, Vasques-Novoa F, Leite-Moreira A. Interplay between worsening kidney function and cardiovascular events in patients with type 2 diabetes: an analysis from the ACCORD trial. BMJ Open Diabetes Res Care. 2021 Jul;9(1):e002408. doi: 10.1136/bmjdrc-2021-002408. PMID 34326100
- [Derived] Kloecker DE, Khunti K, Davies MJ, Pitocco D, Zaccardi F. Microvascular Disease and Risk of Cardiovascular Events and Death From Intensive Treatment in Type 2 Diabetes: The ACCORDION Study. Mayo Clin Proc. 2021 Jun;96(6):1458-1469. doi: 10.1016/j.mayocp.2020.08.047. Epub 2021 May 2. PMID 33952397
- [Derived] Zhou JJ, Koska J, Bahn G, Reaven P. Fasting Glucose Variation Predicts Microvascular Risk in ACCORD and VADT. J Clin Endocrinol Metab. 2021 Mar 25;106(4):1150-1162. doi: 10.1210/clinem/dgaa941. PMID 33367811
- [Derived] Tang Y, Shah H, Bueno Junior CR, Sun X, Mitri J, Sambataro M, Sambado L, Gerstein HC, Fonseca V, Doria A, Pop-Busui R. Intensive Risk Factor Management and Cardiovascular Autonomic Neuropathy in Type 2 Diabetes: The ACCORD Trial. Diabetes Care. 2021 Jan;44(1):164-173. doi: 10.2337/dc20-1842. Epub 2020 Nov 3. PMID 33144354
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Singleton MJ, Soliman EZ, Bertoni AG, Whalen SP, Bhave PD, Yeboah J. Effect of Intensive Glycemic and Blood Pressure Control on QT Prolongation in Diabetes: The ACCORD Trial. Diabetes. 2020 Oct;69(10):2186-2193. doi: 10.2337/db20-0401. Epub 2020 Jul 30. PMID 32732305
- [Derived] Collard D, Brouwer TF, Olde Engberink RHG, Zwinderman AH, Vogt L, van den Born BH. Initial Estimated Glomerular Filtration Rate Decline and Long-Term Renal Function During Intensive Antihypertensive Therapy: A Post Hoc Analysis of the SPRINT and ACCORD-BP Randomized Controlled Trials. Hypertension. 2020 May;75(5):1205-1212. doi: 10.1161/HYPERTENSIONAHA.119.14659. Epub 2020 Mar 30. PMID 32223381
- [Derived] Xing Z, Peng Z, Wang X, Zhu Z, Pei J, Hu X, Chai X. Waist circumference is associated with major adverse cardiovascular events in male but not female patients with type-2 diabetes mellitus. Cardiovasc Diabetol. 2020 Mar 25;19(1):39. doi: 10.1186/s12933-020-01007-6. PMID 32213183
- [Derived] Zhu L, Hayen A, Bell KJL. Legacy effect of fibrate add-on therapy in diabetic patients with dyslipidemia: a secondary analysis of the ACCORDION study. Cardiovasc Diabetol. 2020 Mar 5;19(1):28. doi: 10.1186/s12933-020-01002-x. PMID 32138746
- [Derived] Xing Z, Tang L, Chen J, Pei J, Chen P, Fang Z, Zhou S, Hu X. Association of predicted lean body mass and fat mass with cardiovascular events in patients with type 2 diabetes mellitus. CMAJ. 2019 Sep 23;191(38):E1042-E1048. doi: 10.1503/cmaj.190124. PMID 31548190
- [Derived] Segar MW, Vaduganathan M, Patel KV, McGuire DK, Butler J, Fonarow GC, Basit M, Kannan V, Grodin JL, Everett B, Willett D, Berry J, Pandey A. Machine Learning to Predict the Risk of Incident Heart Failure Hospitalization Among Patients With Diabetes: The WATCH-DM Risk Score. Diabetes Care. 2019 Dec;42(12):2298-2306. doi: 10.2337/dc19-0587. Epub 2019 Sep 13. PMID 31519694
- [Derived] Smith SM, Gurka MJ, Winterstein AG, Pepine CJ, Cooper-DeHoff RM. Incidence, prevalence, and predictors of treatment-resistant hypertension with intensive blood pressure lowering. J Clin Hypertens (Greenwich). 2019 Jun;21(6):825-834. doi: 10.1111/jch.13550. Epub 2019 May 7. PMID 31066177
- [Derived] Duan T, Rajpurkar P, Laird D, Ng AY, Basu S. Clinical Value of Predicting Individual Treatment Effects for Intensive Blood Pressure Therapy. Circ Cardiovasc Qual Outcomes. 2019 Mar;12(3):e005010. doi: 10.1161/CIRCOUTCOMES.118.005010. PMID 30857410
- [Derived] Juraschek SP, Lipsitz LA, Beach JL, Mukamal KJ. Association of Orthostatic Hypotension Timing With Clinical Events in Adults With Diabetes and Hypertension: Results From the ACCORD Trial. Am J Hypertens. 2019 Jun 11;32(7):684-694. doi: 10.1093/ajh/hpz015. PMID 30715100
- [Derived] Collard D, Brouwer TF, Peters RJG, Vogt L, van den Born BH. Creatinine Rise During Blood Pressure Therapy and the Risk of Adverse Clinical Outcomes in Patients With Type 2 Diabetes Mellitus. Hypertension. 2018 Dec;72(6):1337-1344. doi: 10.1161/HYPERTENSIONAHA.118.11944. PMID 30571235
- [Derived] Xing Z, Pei J, Huang J, Peng X, Chen P, Hu X. Relationship of Obesity to Adverse Events Among Patients With Mean 10-Year History of Type 2 Diabetes Mellitus: Results of the ACCORD Study. J Am Heart Assoc. 2018 Nov 20;7(22):e010512. doi: 10.1161/JAHA.118.010512. PMID 30554548
- [Derived] Morieri ML, Gao H, Pigeyre M, Shah HS, Sjaarda J, Mendonca C, Hastings T, Buranasupkajorn P, Motsinger-Reif AA, Rotroff DM, Sigal RJ, Marcovina SM, Kraft P, Buse JB, Wagner MJ, Gerstein HC, Mychaleckyj JC, Pare G, Doria A. Genetic Tools for Coronary Risk Assessment in Type 2 Diabetes: A Cohort Study From the ACCORD Clinical Trial. Diabetes Care. 2018 Nov;41(11):2404-2413. doi: 10.2337/dc18-0709. Epub 2018 Sep 27. PMID 30262460
- [Derived] Beddhu S, Greene T, Boucher R, Cushman WC, Wei G, Stoddard G, Ix JH, Chonchol M, Kramer H, Cheung AK, Kimmel PL, Whelton PK, Chertow GM. Intensive systolic blood pressure control and incident chronic kidney disease in people with and without diabetes mellitus: secondary analyses of two randomised controlled trials. Lancet Diabetes Endocrinol. 2018 Jul;6(7):555-563. doi: 10.1016/S2213-8587(18)30099-8. Epub 2018 Apr 21. PMID 29685860
- [Derived] Brouwer TF, Vehmeijer JT, Kalkman DN, Berger WR, van den Born BH, Peters RJ, Knops RE. Intensive Blood Pressure Lowering in Patients With and Patients Without Type 2 Diabetes: A Pooled Analysis From Two Randomized Trials. Diabetes Care. 2018 Jun;41(6):1142-1148. doi: 10.2337/dc17-1722. Epub 2017 Dec 6. PMID 29212825
- [Derived] Shah HS, Morieri ML, Marcovina SM, Sigal RJ, Gerstein HC, Wagner MJ, Motsinger-Reif AA, Buse JB, Kraft P, Mychaleckyj JC, Doria A. Modulation of GLP-1 Levels by a Genetic Variant That Regulates the Cardiovascular Effects of Intensive Glycemic Control in ACCORD. Diabetes Care. 2018 Feb;41(2):348-355. doi: 10.2337/dc17-1638. Epub 2017 Nov 28. PMID 29183908
- [Derived] Kalkman DN, Brouwer TF, Vehmeijer JT, Berger WR, Knops RE, de Winter RJ, Peters RJ, van den Born BH. J Curve in Patients Randomly Assigned to Different Systolic Blood Pressure Targets: An Experimental Approach to an Observational Paradigm. Circulation. 2017 Dec 5;136(23):2220-2229. doi: 10.1161/CIRCULATIONAHA.117.030342. Epub 2017 Sep 22. PMID 28939617
- [Derived] O Hartaigh B, Szymonifka J, Okin PM. Achieving target SBP for lowering the risk of major adverse cardiovascular events in persons with diabetes mellitus. J Hypertens. 2018 Jan;36(1):101-109. doi: 10.1097/HJH.0000000000001515. PMID 28832365
- [Derived] Elam MB, Ginsberg HN, Lovato LC, Corson M, Largay J, Leiter LA, Lopez C, O'Connor PJ, Sweeney ME, Weiss D, Friedewald WT, Buse JB, Gerstein HC, Probstfield J, Grimm R, Ismail-Beigi F, Goff DC Jr, Fleg JL, Rosenberg Y, Byington RP; ACCORDION Study Investigators. Association of Fenofibrate Therapy With Long-term Cardiovascular Risk in Statin-Treated Patients With Type 2 Diabetes. JAMA Cardiol. 2017 Apr 1;2(4):370-380. doi: 10.1001/jamacardio.2016.4828. PMID 28030716
- [Derived] Murray AM, Hsu FC, Williamson JD, Bryan RN, Gerstein HC, Sullivan MD, Miller ME, Leng I, Lovato LL, Launer LJ; Action to Control Cardiovascular Risk in Diabetes Follow-On Memory in Diabetes (ACCORDION MIND) Investigators. ACCORDION MIND: results of the observational extension of the ACCORD MIND randomised trial. Diabetologia. 2017 Jan;60(1):69-80. doi: 10.1007/s00125-016-4118-x. Epub 2016 Oct 20. PMID 27766347
- [Derived] Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Eye Study Group and the Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Study Group. Persistent Effects of Intensive Glycemic Control on Retinopathy in Type 2 Diabetes in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Follow-On Study. Diabetes Care. 2016 Jul;39(7):1089-100. doi: 10.2337/dc16-0024. Epub 2016 Jun 11. PMID 27289122
- [Derived] Papademetriou V, Zaheer M, Doumas M, Lovato L, Applegate WB, Tsioufis C, Mottle A, Punthakee Z, Cushman WC; ACCORD Study Group. Cardiovascular Outcomes in Action to Control Cardiovascular Risk in Diabetes: Impact of Blood Pressure Level and Presence of Kidney Disease. Am J Nephrol. 2016;43(4):271-80. doi: 10.1159/000446122. Epub 2016 Apr 29. PMID 27161620
- [Derived] ACCORD Study Group. Nine-Year Effects of 3.7 Years of Intensive Glycemic Control on Cardiovascular Outcomes. Diabetes Care. 2016 May;39(5):701-8. doi: 10.2337/dc15-2283. Epub 2016 Jan 28. PMID 26822326
- [Derived] Chen LY, Bigger JT, Hickey KT, Chen H, Lopez-Jimenez C, Banerji MA, Evans G, Fleg JL, Papademetriou V, Thomas A, Woo V, Seaquist ER, Soliman EZ. Effect of Intensive Blood Pressure Lowering on Incident Atrial Fibrillation and P-Wave Indices in the ACCORD Blood Pressure Trial. Am J Hypertens. 2016 Nov 1;29(11):1276-1282. doi: 10.1093/ajh/hpv172. PMID 26476086
- [Derived] Siraj ES, Rubin DJ, Riddle MC, Miller ME, Hsu FC, Ismail-Beigi F, Chen SH, Ambrosius WT, Thomas A, Bestermann W, Buse JB, Genuth S, Joyce C, Kovacs CS, O'Connor PJ, Sigal RJ, Solomon S; ACCORD Investigators. Insulin Dose and Cardiovascular Mortality in the ACCORD Trial. Diabetes Care. 2015 Nov;38(11):2000-8. doi: 10.2337/dc15-0598. Epub 2015 Oct 13. PMID 26464212
- [Derived] Soliman EZ, Byington RP, Bigger JT, Evans G, Okin PM, Goff DC Jr, Chen H. Effect of Intensive Blood Pressure Lowering on Left Ventricular Hypertrophy in Patients With Diabetes Mellitus: Action to Control Cardiovascular Risk in Diabetes Blood Pressure Trial. Hypertension. 2015 Dec;66(6):1123-9. doi: 10.1161/HYPERTENSIONAHA.115.06236. Epub 2015 Oct 12. PMID 26459421
- [Derived] Chow LS, Chen H, Miller ME, Marcovina SM, Seaquist ER. Biomarkers associated with severe hypoglycaemia and death in ACCORD. Diabet Med. 2016 Aug;33(8):1076-83. doi: 10.1111/dme.12883. Epub 2015 Sep 6. PMID 26261902
- [Derived] Hempe JM, Liu S, Myers L, McCarter RJ, Buse JB, Fonseca V. The hemoglobin glycation index identifies subpopulations with harms or benefits from intensive treatment in the ACCORD trial. Diabetes Care. 2015 Jun;38(6):1067-74. doi: 10.2337/dc14-1844. Epub 2015 Apr 17. PMID 25887355
- [Derived] Espeland MA, Probstfield J, Hire D, Redmon JB, Evans GW, Coday M, Lewis CE, Johnson KC, Wilmoth S, Bahnson J, Dulin MF, Green JB, Knowler WC, Kitabchi A, Murillo AL, Osei K, Rehman SU, Cushman WC; Look AHEAD Research Group; ACCORD Study Group. Systolic Blood Pressure Control Among Individuals With Type 2 Diabetes: A Comparative Effectiveness Analysis of Three Interventions. Am J Hypertens. 2015 Aug;28(8):995-1009. doi: 10.1093/ajh/hpu292. Epub 2015 Feb 9. PMID 25666468
- [Derived] Chow LS, Chen H, Miller ME, Marcovina SM, Seaquist ER. Biomarkers related to severe hypoglycaemia and lack of good glycaemic control in ACCORD. Diabetologia. 2015 Jun;58(6):1160-6. doi: 10.1007/s00125-015-3512-0. Epub 2015 Feb 5. PMID 25652389
- [Derived] Zhang Z, Lovato J, Battapady H, Davatzikos C, Gerstein HC, Ismail-Beigi F, Launer LJ, Murray A, Punthakee Z, Tirado AA, Williamson J, Bryan RN, Miller ME. Effect of hypoglycemia on brain structure in people with type 2 diabetes: epidemiological analysis of the ACCORD-MIND MRI trial. Diabetes Care. 2014 Dec;37(12):3279-85. doi: 10.2337/dc14-0973. Epub 2014 Sep 29. PMID 25267796
- [Derived] Papademetriou V, Lovato L, Doumas M, Nylen E, Mottl A, Cohen RM, Applegate WB, Puntakee Z, Yale JF, Cushman WC; ACCORD Study Group. Chronic kidney disease and intensive glycemic control increase cardiovascular risk in patients with type 2 diabetes. Kidney Int. 2015 Mar;87(3):649-59. doi: 10.1038/ki.2014.296. Epub 2014 Sep 17. PMID 25229335
- [Derived] Hugenschmidt CE, Lovato JF, Ambrosius WT, Bryan RN, Gerstein HC, Horowitz KR, Launer LJ, Lazar RM, Murray AM, Chew EY, Danis RP, Williamson JD, Miller ME, Ding J. The cross-sectional and longitudinal associations of diabetic retinopathy with cognitive function and brain MRI findings: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Diabetes Care. 2014 Dec;37(12):3244-52. doi: 10.2337/dc14-0502. Epub 2014 Sep 5. PMID 25193529
- [Derived] Chew EY, Davis MD, Danis RP, Lovato JF, Perdue LH, Greven C, Genuth S, Goff DC, Leiter LA, Ismail-Beigi F, Ambrosius WT; Action to Control Cardiovascular Risk in Diabetes Eye Study Research Group. The effects of medical management on the progression of diabetic retinopathy in persons with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study. Ophthalmology. 2014 Dec;121(12):2443-51. doi: 10.1016/j.ophtha.2014.07.019. Epub 2014 Aug 29. PMID 25172198
- [Derived] Fatemi O, Yuriditsky E, Tsioufis C, Tsachris D, Morgan T, Basile J, Bigger T, Cushman W, Goff D, Soliman EZ, Thomas A, Papademetriou V. Impact of intensive glycemic control on the incidence of atrial fibrillation and associated cardiovascular outcomes in patients with type 2 diabetes mellitus (from the Action to Control Cardiovascular Risk in Diabetes Study). Am J Cardiol. 2014 Oct 15;114(8):1217-22. doi: 10.1016/j.amjcard.2014.07.045. Epub 2014 Jul 30. PMID 25159234
- [Derived] Margolis KL, Palermo L, Vittinghoff E, Evans GW, Atkinson HH, Hamilton BP, Josse RG, O'Connor PJ, Simmons DL, Tiktin M, Schwartz AV. Intensive blood pressure control, falls, and fractures in patients with type 2 diabetes: the ACCORD trial. J Gen Intern Med. 2014 Dec;29(12):1599-606. doi: 10.1007/s11606-014-2961-3. Epub 2014 Aug 16. PMID 25127725
- [Derived] Gerstein HC, Miller ME, Ismail-Beigi F, Largay J, McDonald C, Lochnan HA, Booth GL; ACCORD Study Group. Effects of intensive glycaemic control on ischaemic heart disease: analysis of data from the randomised, controlled ACCORD trial. Lancet. 2014 Nov 29;384(9958):1936-41. doi: 10.1016/S0140-6736(14)60611-5. Epub 2014 Jul 31. PMID 25088437
- [Derived] Bryan RN, Bilello M, Davatzikos C, Lazar RM, Murray A, Horowitz K, Lovato J, Miller ME, Williamson J, Launer LJ. Effect of diabetes on brain structure: the action to control cardiovascular risk in diabetes MR imaging baseline data. Radiology. 2014 Jul;272(1):210-6. doi: 10.1148/radiol.14131494. Epub 2014 Apr 29. PMID 24779562
- [Derived] Margolis KL, O'Connor PJ, Morgan TM, Buse JB, Cohen RM, Cushman WC, Cutler JA, Evans GW, Gerstein HC, Grimm RH Jr, Lipkin EW, Narayan KM, Riddle MC Jr, Sood A, Goff DC Jr. Outcomes of combined cardiovascular risk factor management strategies in type 2 diabetes: the ACCORD randomized trial. Diabetes Care. 2014 Jun;37(6):1721-8. doi: 10.2337/dc13-2334. Epub 2014 Mar 4. PMID 24595629
- [Derived] Williamson JD, Launer LJ, Bryan RN, Coker LH, Lazar RM, Gerstein HC, Murray AM, Sullivan MD, Horowitz KR, Ding J, Marcovina S, Lovato L, Lovato J, Margolis KL, Davatzikos C, Barzilay J, Ginsberg HN, Linz PE, Miller ME; Action to Control Cardiovascular Risk in Diabetes Memory in Diabetes Investigators. Cognitive function and brain structure in persons with type 2 diabetes mellitus after intensive lowering of blood pressure and lipid levels: a randomized clinical trial. JAMA Intern Med. 2014 Mar;174(3):324-33. doi: 10.1001/jamainternmed.2013.13656. PMID 24493100
- [Derived] Linz PE, Lovato LC, Byington RP, O'Connor PJ, Leiter LA, Weiss D, Force RW, Crouse JR, Ismail-Beigi F, Simmons DL, Papademetriou V, Ginsberg HN, Elam MB. Paradoxical reduction in HDL-C with fenofibrate and thiazolidinedione therapy in type 2 diabetes: the ACCORD Lipid Trial. Diabetes Care. 2014;37(3):686-93. doi: 10.2337/dc13-0790. Epub 2013 Dec 2. PMID 24296848
- [Derived] Miller ME, Williamson JD, Gerstein HC, Byington RP, Cushman WC, Ginsberg HN, Ambrosius WT, Lovato L, Applegate WB; ACCORD Investigators. Effects of randomization to intensive glucose control on adverse events, cardiovascular disease, and mortality in older versus younger adults in the ACCORD Trial. Diabetes Care. 2014;37(3):634-43. doi: 10.2337/dc13-1545. Epub 2013 Oct 29. PMID 24170759
- [Derived] Barzilay JI, Lovato JF, Murray AM, Williamson J, Ismail-Beigi F, Karl D, Papademetriou V, Launer LJ. Albuminuria and cognitive decline in people with diabetes and normal renal function. Clin J Am Soc Nephrol. 2013 Nov;8(11):1907-14. doi: 10.2215/CJN.11321112. Epub 2013 Aug 29. PMID 23990163
- [Derived] Fonseca V, McDuffie R, Calles J, Cohen RM, Feeney P, Feinglos M, Gerstein HC, Ismail-Beigi F, Morgan TM, Pop-Busui R, Riddle MC; ACCORD Study Group. Determinants of weight gain in the action to control cardiovascular risk in diabetes trial. Diabetes Care. 2013 Aug;36(8):2162-8. doi: 10.2337/dc12-1391. Epub 2013 Feb 14. PMID 23412077
- [Derived] Gerstein HC, Ambrosius WT, Danis R, Ismail-Beigi F, Cushman W, Calles J, Banerji M, Schubart U, Chew EY; ACCORD Study Group. Diabetic retinopathy, its progression, and incident cardiovascular events in the ACCORD trial. Diabetes Care. 2013 May;36(5):1266-71. doi: 10.2337/dc12-1311. Epub 2012 Dec 13. PMID 23238658
- [Derived] Reyes-Soffer G, Ngai CI, Lovato L, Karmally W, Ramakrishnan R, Holleran S, Ginsberg HN. Effect of combination therapy with fenofibrate and simvastatin on postprandial lipemia in the ACCORD lipid trial. Diabetes Care. 2013 Feb;36(2):422-8. doi: 10.2337/dc11-2556. Epub 2012 Oct 1. PMID 23033246
- [Derived] Barzilay JI, Howard AG, Evans GW, Fleg JL, Cohen RM, Booth GL, Kimel AR, Pedley CF, Cushman WC. Intensive blood pressure treatment does not improve cardiovascular outcomes in centrally obese hypertensive individuals with diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Blood Pressure Trial. Diabetes Care. 2012 Jul;35(7):1401-5. doi: 10.2337/dc11-1827. PMID 22723577
- [Derived] Bonds DE, Miller ME, Dudl J, Feinglos M, Ismail-Beigi F, Malozowski S, Seaquist E, Simmons DL, Sood A. Severe hypoglycemia symptoms, antecedent behaviors, immediate consequences and association with glycemia medication usage: Secondary analysis of the ACCORD clinical trial data. BMC Endocr Disord. 2012 May 30;12:5. doi: 10.1186/1472-6823-12-5. PMID 22646230
- [Derived] Sullivan MD, O'Connor P, Feeney P, Hire D, Simmons DL, Raisch DW, Fine LJ, Narayan KM, Ali MK, Katon WJ. Depression predicts all-cause mortality: epidemiological evaluation from the ACCORD HRQL substudy. Diabetes Care. 2012 Aug;35(8):1708-15. doi: 10.2337/dc11-1791. Epub 2012 May 22. PMID 22619083
- [Derived] Raisch DW, Feeney P, Goff DC Jr, Narayan KM, O'Connor PJ, Zhang P, Hire DG, Sullivan MD. Baseline comparison of three health utility measures and the feeling thermometer among participants in the Action to Control Cardiovascular Risk in Diabetes trial. Cardiovasc Diabetol. 2012 Jul 11;11:35. doi: 10.1186/1475-2840-11-35. PMID 22515638
- [Derived] Bonds DE, Craven TE, Buse J, Crouse JR, Cuddihy R, Elam M, Ginsberg HN, Kirchner K, Marcovina S, Mychaleckyj JC, O'Connor PJ, Sperl-Hillen JA. Fenofibrate-associated changes in renal function and relationship to clinical outcomes among individuals with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) experience. Diabetologia. 2012 Jun;55(6):1641-50. doi: 10.1007/s00125-012-2524-2. Epub 2012 Mar 27. PMID 22450889
- [Derived] Mychaleckyj JC, Craven T, Nayak U, Buse J, Crouse JR, Elam M, Kirchner K, Lorber D, Marcovina S, Sivitz W, Sperl-Hillen J, Bonds DE, Ginsberg HN. Reversibility of fenofibrate therapy-induced renal function impairment in ACCORD type 2 diabetic participants. Diabetes Care. 2012 May;35(5):1008-14. doi: 10.2337/dc11-1811. Epub 2012 Mar 19. PMID 22432114
- [Derived] Punthakee Z, Miller ME, Launer LJ, Williamson JD, Lazar RM, Cukierman-Yaffee T, Seaquist ER, Ismail-Beigi F, Sullivan MD, Lovato LC, Bergenstal RM, Gerstein HC; ACCORD Group of Investigators; ACCORD-MIND Investigators. Poor cognitive function and risk of severe hypoglycemia in type 2 diabetes: post hoc epidemiologic analysis of the ACCORD trial. Diabetes Care. 2012 Apr;35(4):787-93. doi: 10.2337/dc11-1855. Epub 2012 Feb 28. PMID 22374637
- [Derived] Seaquist ER, Miller ME, Bonds DE, Feinglos M, Goff DC Jr, Peterson K, Senior P; ACCORD Investigators. The impact of frequent and unrecognized hypoglycemia on mortality in the ACCORD study. Diabetes Care. 2012 Feb;35(2):409-14. doi: 10.2337/dc11-0996. Epub 2011 Dec 16. PMID 22179956
- [Derived] Genuth S, Ismail-Beigi F. Clinical implications of the ACCORD trial. J Clin Endocrinol Metab. 2012 Jan;97(1):41-8. doi: 10.1210/jc.2011-1679. Epub 2011 Nov 2. PMID 22049171
- [Derived] Samaropoulos XF, Light L, Ambrosius WT, Marcovina SM, Probstfield J, Goff DC Jr. The effect of intensive risk factor management in type 2 diabetes on inflammatory biomarkers. Diabetes Res Clin Pract. 2012 Mar;95(3):389-98. doi: 10.1016/j.diabres.2011.09.027. Epub 2011 Oct 22. PMID 22019270
- [Derived] Launer LJ, Miller ME, Williamson JD, Lazar RM, Gerstein HC, Murray AM, Sullivan M, Horowitz KR, Ding J, Marcovina S, Lovato LC, Lovato J, Margolis KL, O'Connor P, Lipkin EW, Hirsch J, Coker L, Maldjian J, Sunshine JL, Truwit C, Davatzikos C, Bryan RN; ACCORD MIND investigators. Effects of intensive glucose lowering on brain structure and function in people with type 2 diabetes (ACCORD MIND): a randomised open-label substudy. Lancet Neurol. 2011 Nov;10(11):969-77. doi: 10.1016/S1474-4422(11)70188-0. Epub 2011 Sep 28. PMID 21958949
- [Derived] Mychaleckyj JC, Farber EA, Chmielewski J, Artale J, Light LS, Bowden DW, Hou X, Marcovina SM. Buffy coat specimens remain viable as a DNA source for highly multiplexed genome-wide genetic tests after long term storage. J Transl Med. 2011 Jun 10;9:91. doi: 10.1186/1479-5876-9-91. PMID 21663644
- [Derived] ACCORD Study Group; Gerstein HC, Miller ME, Genuth S, Ismail-Beigi F, Buse JB, Goff DC Jr, Probstfield JL, Cushman WC, Ginsberg HN, Bigger JT, Grimm RH Jr, Byington RP, Rosenberg YD, Friedewald WT. Long-term effects of intensive glucose lowering on cardiovascular outcomes. N Engl J Med. 2011 Mar 3;364(9):818-28. doi: 10.1056/NEJMoa1006524. PMID 21366473
- [Derived] Ismail-Beigi F, Craven T, Banerji MA, Basile J, Calles J, Cohen RM, Cuddihy R, Cushman WC, Genuth S, Grimm RH Jr, Hamilton BP, Hoogwerf B, Karl D, Katz L, Krikorian A, O'Connor P, Pop-Busui R, Schubart U, Simmons D, Taylor H, Thomas A, Weiss D, Hramiak I; ACCORD trial group. Effect of intensive treatment of hyperglycaemia on microvascular outcomes in type 2 diabetes: an analysis of the ACCORD randomised trial. Lancet. 2010 Aug 7;376(9739):419-30. doi: 10.1016/S0140-6736(10)60576-4. Epub 2010 Jun 30. PMID 20594588
- [Derived] ACCORD Study Group; ACCORD Eye Study Group; Chew EY, Ambrosius WT, Davis MD, Danis RP, Gangaputra S, Greven CM, Hubbard L, Esser BA, Lovato JF, Perdue LH, Goff DC Jr, Cushman WC, Ginsberg HN, Elam MB, Genuth S, Gerstein HC, Schubart U, Fine LJ. Effects of medical therapies on retinopathy progression in type 2 diabetes. N Engl J Med. 2010 Jul 15;363(3):233-44. doi: 10.1056/NEJMoa1001288. Epub 2010 Jun 29. PMID 20587587
- [Derived] Strylewicz G, Doctor J. Evaluation of an automated method to assist with error detection in the ACCORD central laboratory. Clin Trials. 2010 Aug;7(4):380-9. doi: 10.1177/1740774510372779. Epub 2010 Jun 22. PMID 20571135
- [Derived] Riddle MC, Ambrosius WT, Brillon DJ, Buse JB, Byington RP, Cohen RM, Goff DC Jr, Malozowski S, Margolis KL, Probstfield JL, Schnall A, Seaquist ER; Action to Control Cardiovascular Risk in Diabetes Investigators. Epidemiologic relationships between A1C and all-cause mortality during a median 3.4-year follow-up of glycemic treatment in the ACCORD trial. Diabetes Care. 2010 May;33(5):983-90. doi: 10.2337/dc09-1278. PMID 20427682
- [Derived] ACCORD Study Group; Ginsberg HN, Elam MB, Lovato LC, Crouse JR 3rd, Leiter LA, Linz P, Friedewald WT, Buse JB, Gerstein HC, Probstfield J, Grimm RH, Ismail-Beigi F, Bigger JT, Goff DC Jr, Cushman WC, Simons-Morton DG, Byington RP. Effects of combination lipid therapy in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1563-74. doi: 10.1056/NEJMoa1001282. Epub 2010 Mar 14. PMID 20228404
- [Derived] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Derived] Pop-Busui R, Evans GW, Gerstein HC, Fonseca V, Fleg JL, Hoogwerf BJ, Genuth S, Grimm RH, Corson MA, Prineas R; Action to Control Cardiovascular Risk in Diabetes Study Group. Effects of cardiac autonomic dysfunction on mortality risk in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial. Diabetes Care. 2010 Jul;33(7):1578-84. doi: 10.2337/dc10-0125. Epub 2010 Mar 9. PMID 20215456
- [Derived] Miller ME, Bonds DE, Gerstein HC, Seaquist ER, Bergenstal RM, Calles-Escandon J, Childress RD, Craven TE, Cuddihy RM, Dailey G, Feinglos MN, Ismail-Beigi F, Largay JF, O'Connor PJ, Paul T, Savage PJ, Schubart UK, Sood A, Genuth S; ACCORD Investigators. The effects of baseline characteristics, glycaemia treatment approach, and glycated haemoglobin concentration on the risk of severe hypoglycaemia: post hoc epidemiological analysis of the ACCORD study. BMJ. 2010 Jan 8;340:b5444. doi: 10.1136/bmj.b5444. PMID 20061360
- [Derived] Bonds DE, Miller ME, Bergenstal RM, Buse JB, Byington RP, Cutler JA, Dudl RJ, Ismail-Beigi F, Kimel AR, Hoogwerf B, Horowitz KR, Savage PJ, Seaquist ER, Simmons DL, Sivitz WI, Speril-Hillen JM, Sweeney ME. The association between symptomatic, severe hypoglycaemia and mortality in type 2 diabetes: retrospective epidemiological analysis of the ACCORD study. BMJ. 2010 Jan 8;340:b4909. doi: 10.1136/bmj.b4909. PMID 20061358
- [Derived] Meier M, Hummel M. Cardiovascular disease and intensive glucose control in type 2 diabetes mellitus: moving practice toward evidence-based strategies. Vasc Health Risk Manag. 2009;5:859-71. doi: 10.2147/vhrm.s4808. Epub 2009 Nov 2. PMID 19898642
- See also: Click here for the ACCORD trial web site — http://www.accordtrial.org/
- Available data/document: Individual Participant Data Set: ACCORD — http://biolincc.nhlbi.nih.gov/studies/accord — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/accord
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/accord
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/accord

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants had established type 2 diabetes and were recruited from 77 clinical centers in the United States (64 sites) and Canada (13 sites). Recruitment occurred in two phases, from January to June 2001 and from February 2003 to October 2005.
Pre-assignment Details: Eligible participants provided evidence of ability to routinely monitor capillary blood sugars from written records or electronic downloads from a self-monitoring blood glucose device (SMBG), or (in cases where such records could not be provided) underwent a 2 to 4-week pre-randomization run-in period to evaluate compliance with SMBG monitoring.
Groups:
- Glycemia Trial: Intensive Control/BP Trial: Intensive Control: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  BP Trial - Open label administration of anti-hypertensive agents to reduce and maintain systolic blood pressure (SBP) level to <120 mmHg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals.
- Glycemia Trial: Intensive Control/BP Trial: Standard Control: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  BP Trial - Open label administration of multiple anti-hypertensive agents to maintain SBP level <140 mm Hg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals.
- Glycemia Trial: Intensive Control/Lipid Trial: Fenofibrate: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  Lipid Trial - Double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 in combination with open label simvastatin. Blinded fenofibrate or placebo plus simvastatin includes double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 or matching placebo in combination with open label simvastatin 20 - 40 mg/day.
- Glycemia Trial: Intensive Control/Lipid Trial: Placebo: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  Double blind administration of placebo matching either 160 mg/day in participants with eGFR ≥50 mL/min/1.73m2 or 54 mg/day in participants with eGFR <50 mL/min/1.73m^2 in combination with open label simvastatin. Blinded fenofibrate or placebo plus simvastatin includes double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 or matching placebo in combination with open label simvastatin 20 - 40 mg/day.
- Glycemia Trial: Standard Control/BP Trial: Intensive Control: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 to 7.9%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  BP Trial - Open label administration of anti-hypertensive agents to reduce and maintain systolic blood pressure (SBP) level to <120 mmHg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals.
- Glycemia Trial: Standard Control/BP Trial: Standard Control: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 to 7.9%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  BP Trial - Open label administration of multiple anti-hypertensive agents to maintain SBP level <140 mm Hg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals (intensive control <120 mm Hg; standard control <140 mm Hg).
- Glycemia Trial: Standard Control/Lipid Trial: Fenofibrate: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 to 7.9%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  Lipid Trial - Double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 in combination with open label simvastatin. Blinded fenofibrate or placebo plus simvastatin includes double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 or matching placebo in combination with open label simvastatin 20 - 40 mg/day.
- Glycemia Trial: Standard Control/Lipid Trial: Placebo: Glycemia Trial - Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 to 7.9%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
  Double blind administration of placebo matching either 160 mg/day in participants with eGFR ≥50 mL/min/1.73m2 or 54 mg/day in participants with eGFR <50 mL/min/1.73m^2 in combination with open label simvastatin. Blinded fenofibrate or placebo plus simvastatin includes double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2 or matching placebo in combination with open label simvastatin 20 - 40 mg/day.
Period: Overall Study
Arm/Group | Glycemia Trial: Intensive Control/BP Trial: Intensive Control | Glycemia Trial: Intensive Control/BP Trial: Standard Control | Glycemia Trial: Intensive Control/Lipid Trial: Fenofibrate | Glycemia Trial: Intensive Control/Lipid Trial: Placebo | Glycemia Trial: Standard Control/BP Trial: Intensive Control | Glycemia Trial: Standard Control/BP Trial: Standard Control | Glycemia Trial: Standard Control/Lipid Trial: Fenofibrate | Glycemia Trial: Standard Control/Lipid Trial: Placebo
Started | 1178 | 1193 | 1374 | 1383 | 1184 | 1178 | 1391 | 1370
Completed | 1016 | 1057 | 1204 | 1205 | 1049 | 1026 | 1242 | 1224
Not Completed | 162 | 136 | 170 | 178 | 135 | 152 | 149 | 146
Not completed — Death | 86 | 67 | 112 | 126 | 64 | 77 | 91 | 95
Not completed — Lost to Follow-up | 14 | 14 | 14 | 14 | 15 | 15 | 13 | 14
Not completed — Withdrawal by Subject | 40 | 27 | 28 | 27 | 30 | 32 | 32 | 21
Not completed — missed closeout visit | 22 | 28 | 16 | 11 | 26 | 28 | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Glycemia Trial: Intensive Control: Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels <6.0%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
- Glycemia Trial: Standard Control: Open label administration of oral anti-hyperglycemic agents and/or insulin in combination with dietary/lifestyle advice as needed to achieve glycated hemoglobin (HbA1c) levels of 7.0 to 7.9%. Anti-hyperglycemic agents include multiple drugs including insulins and oral anti-hyperglycemic agents as needed to reach Glycemia Trial arm-specific goals.
- Total: Total of all reporting groups
Arm/Group | Glycemia Trial: Intensive Control | Glycemia Trial: Standard Control | Total
Number analyzed (Participants) | 5128 | 5123 | 10251
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (6.8) | 62.2 (6.8) | 62.2 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 1983 | 1969 | 3952
  Male | 3145 | 3154 | 6299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 358 | 379 | 737
  Not Hispanic or Latino | 4770 | 4744 | 9514
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Nonwhite | 1828 | 1819 | 3647
  White | 3300 | 3304 | 6604
Region of Enrollment [Number; unit: participants]
  United States | 4376 | 4367 | 8743
  Canada | 752 | 756 | 1508
Previous cardiovascular disease (CVD) event [Number; unit: participants]
  History of CVD event | 1827 | 1782 | 3609
  No history of CVD event | 3301 | 3341 | 6642
Glycated hemoglobin [Mean (Standard Deviation); unit: percent] | 8.3 (1.1) | 8.3 (1.1) | 8.3 (1.1)
Blood pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic | 136.2 (17.0) | 136.5 (17.2) | 136.4 (17.1)
  Diastolic | 74.8 (10.6) | 75.0 (10.7) | 74.9 (10.7)
Cholesterol [Mean (Standard Deviation); unit: mg/dL]
  LDL | 104.9 (34.0) | 104.9 (33.8) | 104.9 (33.9)
  HDL | 41.8 (11.8) | 41.9 (11.5) | 41.9 (11.6)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 156 [105 to 230] | 154 [108 to 226] | 155 [106 to 228]
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 10 [5 to 15] | 10 [5 to 15] | 10 [5 to 15]

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of a Major Cardiovascular Event (MCE); Specifically Nonfatal Heart Attack, Nonfatal Stroke, or Cardiovascular Death (Measured Throughout the Study) in the Glycemia Trial.
Description: Time to first occurrence of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death. This was the primary outcome measure in all three trials: Glycemia (all participants), Blood Pressure (subgroup of participants not in Lipid Trial), and Lipid (subgroup of participants not in Blood Pressure Trial).
  In the Glycemia Trial, a finding of higher mortality in the intensive arm group led to an early discontinuation of therapy after a mean of 3.5 years of follow-up. Intensive arm participants were transitioned to standard arm strategy over a period of 0.2 year and followed for an additional 1.2 years to the planned end of the Glycemia Trial while participating in one of the other sub-trials (BP or Lipid) to their planned completion.
Time Frame: 4.9 years
Population: The population analyzed included all participants randomized and was performed by intention to treat with right-censoring of participants who did not complete follow-up prior to occurrence of MCE.
Measure: Number; unit: participants
Arm/Group | Glycemia Trial: Intensive Control | Glycemia Trial: Standard Control
Number analyzed (Participants) | 5128 | 5123
participants | 503 | 543
Statistical Analysis 1: Comparison: Glycemia Trial: Intensive Control vs Glycemia Trial: Standard Control; Adjustment performed for the following pre-specified factors: sub-trial assignment (Blood Pressure Trial or Lipid Trial), assignment to intensive BP group in BP Trial, assignment to fenofibrate group in Lipid Trial, the seven clinical center networks, and presence of clinical cardiovascular disease at baseline; Test type: Superiority or Other; p = 0.12, Regression, Cox — P-value presented is not adjusted for multiple comparisons. A priori significance level was 0.05; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.81 to 1.03]

2. Secondary Outcome: Death From Any Cause in the Glycemia Trial.
Description: Time to death from any cause. Secondary measure for Glycemia Trial.
  A finding of higher mortality in the intensive-therapy group led to an early discontinuation of therapy after a mean of 3.5 years of follow-up. Intensive arm participants were transitioned to standard arm strategy over a period of 0.2 year and followed for an additional 1.2 years to the planned end of the Glycemia Trial while participating in one of the other sub-trials (BP or Lipid).
Time Frame: 4.9 years
Population: The population analyzed included all participants randomized and was performed by intention to treat with right-censoring of participants who did not complete follow-up prior to death.
Measure: Number; unit: participants
Arm/Group | Glycemia Trial: Intensive Control | Glycemia Trial: Standard Control
Number analyzed (Participants) | 5128 | 5123
participants | 391 | 327
Statistical Analysis 1: Comparison: Glycemia Trial: Intensive Control vs Glycemia Trial: Standard Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.02, Regression, Cox — P-value presented is not adjusted for multiple comparisons. A priori significance level was 0.05; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [1.03 to 1.38]

3. Primary Outcome: First Occurrence of Major Cardiovascular Event (MCE) in the Blood Pressure Trial.
Description: Time to first occurrence of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death. Primary outcome for Blood Pressure Trial.
Time Frame: 4.7 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- BP Trial: Intensive Control: Open label administration of anti-hypertensive agents to reduce and maintain systolic blood pressure (SBP) level to <120 mmHg. Anti-hypertensive agents include multiple anti-hypertensive agents as needed to reach Blood Pressure Trial arm-specific goals.
- BP Trial: Standard Control: Open label administration of multiple anti-hypertensive agents to maintain SBP level <140 mm Hg. Anti-hypertensive agents multiple anti-hypertensive agents as needed to reach Blood Pressure Trial arm-specific goals.
Arm/Group | BP Trial: Intensive Control | BP Trial: Standard Control
Number analyzed (Participants) | 2363 | 2371
participants | 208 | 237
Statistical Analysis 1: Comparison: BP Trial: Intensive Control vs BP Trial: Standard Control; Recruitment for the Blood PressureTrial was designed to enroll 4200 participant to have 94% power to detect a 20% reduction in the rate of MCE for patients in the intensive-therapy group as compared with the standard-therapy group, assuming a two-sided alpha level of 0.05, a primary-outcome rate of 4% per year in the standard-therapy group, and a planned average follow-up of approximately 5.6 years; Test type: Superiority or Other; p = 0.20, Regression, Cox — P-value is adjusted for interim monitoring. A priori significance level was 0.05; Adjustment for the seven clinical center networks and presence of clinical cardiovascular disease at baseline as pre-specified in the study protocol; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.06]

4. Secondary Outcome: Stroke in the Blood Pressure Trial.
Description: Time to first occurrence of nonfatal or fatal stroke among participants in the BP Trial.
Time Frame: 4.7 years
Population: The population analyzed included all participants randomized and was performed by intention to treat with right-censoring of participants who did not complete follow-up prior to occurrence of stroke.
Measure: Number; unit: participants
Groups:
- BP Trial: Intensive Control: Open label administration of anti-hypertensive agents to reduce and maintain systolic blood pressure (SBP) level to <120 mmHg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals.
- BP Trial: Standard Control: Open label administration of multiple anti-hypertensive agents to maintain SBP level to <140 mm Hg. Anti-hypertensive agents include multiple anti-hypertensive medications as needed to reach Blood Pressure Trial arm-specific goals.
Arm/Group | BP Trial: Intensive Control | BP Trial: Standard Control
Number analyzed (Participants) | 2363 | 2371
participants | 36 | 62
Statistical Analysis 1: Comparison: BP Trial: Intensive Control vs BP Trial: Standard Control; Test type: Superiority or Other; p = 0.01, Regression, Cox — P-value presented is not adjusted for multiple comparisons. A priori significance level was 0.05; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.39 to 0.89]

5. Primary Outcome: First Occurrence of Major Cardiovascular Event (MCE) in the Lipid Trial.
Description: Time to first occurrence of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death in Lipid Trial participants.
Time Frame: 4.7 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Lipid Trial: Fenofibrate: Double blind administration of 160 mg/day of fenofibrate in participants with estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m^2 or 54 mg/day in patients with eGFR <50 mL/min/1.73m^2, in combination with open label simvastatin 20 - 40 mg/day.
- Lipid Trial: Placebo: Double blind administration of placebo matching either 160 mg/day in participants with eGFR ≥50 mL/min/1.73m^2 or 54 mg/day in participants with eGFR <50 mL/min/1.73m^2, in combination with open label simvastatin 20 - 40 mg/day.
Arm/Group | Lipid Trial: Fenofibrate | Lipid Trial: Placebo
Number analyzed (Participants) | 2765 | 2753
participants | 291 | 310
Statistical Analysis 1: Comparison: Lipid Trial: Fenofibrate vs Lipid Trial: Placebo; Recruitment for the Glycemia Trial was designed to enroll 5800 participant to have 87% power to detect a 20% reduction in the rate of MCE for patients in the fenofibrate group as compared with the placebo group, assuming a two-sided alpha level of 0.05, a primary-outcome rate of 2.4% per year in the placebo group, and a planned average follow-up of approximately 5.6 years; Test type: Superiority or Other; p = 0.32, Regression, Cox — P-value is adjusted for interim monitoring. A priori significance level was 0.05; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.79 to 1.08]

6. Secondary Outcome: First Occurrence of MCE or Revascularization or Hospitalization for Congestive Heart Failure (CHF) in Lipid Trial.
Description: Time to first occurrence of nonfatal myocardial infarction, nonfatal stroke, cardiovascular death, revascularization procedure or hospitalization for CHF in Lipid Trial participants.
Time Frame: 4.7 years
Population: The population analyzed included all participants randomized and was performed by intention to treat with right-censoring of participants who did not complete follow-up prior occurrence of event.
Measure: Number; unit: participants
Arm/Group | Lipid Trial: Fenofibrate | Lipid Trial: Placebo
Number analyzed (Participants) | 2765 | 2753
participants | 641 | 667
Statistical Analysis 1: Comparison: Lipid Trial: Fenofibrate vs Lipid Trial: Placebo; Test type: Superiority or Other; p = 0.30, Regression, Cox — P-value presented is not adjusted for multiple comparisons. A priori significance level was 0.05; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.85 to 1.05]

ADVERSE EVENTS:
Time Frame: Includes Serious Adverse Events (SAEs) reported after randomization and throughout the planned observation period, mean follow-up was 4.9 years. Data on other (non-serious) adverse events were not collected.
Description: SAEs were defined as any adverse experience that was significantly life threatening and/or resulted in death, permanent disability, hospitalization or prolongation of hospitalization, myositis/myopathy, or hepatitis and were considered by the investigators to be possibly, probably, or definitely related to study treatments.
Arm/Group | Glycemia Trial: Intensive Control | Glycemia Trial: Standard Control
Serious Adverse Events (participants affected / at risk) | 137/5128 | 107/5123
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycemia Trial: Intensive Control (N=5128) | Glycemia Trial: Standard Control (N=5123)
Congestive heart failure (Cardiac disorders) | 34 | 12
Bradycardia, tachycardia, atrial fibrillation (Cardiac disorders) | 13 | 4
Angina/chest pain (Cardiac disorders) | 4 | 5
Myocardial infarction (Cardiac disorders) | 4 | 5
Dizziness, hypotension, syncope (Vascular disorders) | 19 | 17
Edema (Vascular disorders) | 3 | 1
Cerebrovacular accident (Vascular disorders) | 1 | 1
Cholecystitis (Gastrointestinal disorders) | 5 | 11
Hepatitis/liver failure (Gastrointestinal disorders) | 2 | 3
Elevated creatinine, hyponatremia (Gastrointestinal disorders) | 2 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Endocrine disorders) | 5 | 8
Ketoacidosis (Endocrine disorders) | 1 | 0
Hypoglycemia (fatal) (Endocrine disorders) | 0 | 1
Acute or chronic renal failure (Renal and urinary disorders) | 8 | 6
Angioedema (Immune system disorders) | 9 | 4
Thrombocytopenia (Immune system disorders) | 2 | 0
Blood dyscrasia (Immune system disorders) | 1 | 0
Felodipine toxicity (Immune system disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 3
Rhabdomyolisis (Musculoskeletal and connective tissue disorders) | 1 | 2
Fractures (Musculoskeletal and connective tissue disorders) | 1 | 2
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Macular edema (Eye disorders) | 1 | 1
Blurred vision (Eye disorders) | 1 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Motor vehicle accident (fatal) (Injury, poisoning and procedural complications) | 3 | 2
Hyperkalemia (General disorders) | 6 | 5
Hyponatremia (General disorders) | 0 | 4
Severe fluid retention (General disorders) | 3 | 1
Dehydration (General disorders) | 1 | 2
Vertigo (General disorders) | 0 | 1
Anemia (General disorders) | 0 | 1
Hypomagnesemia (General disorders) | 0 | 1
Hyperosmolar nonketotic coma (General disorders) | 1 | 0
Toxic metabolic enecphalopathy (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No